CLINICAL TRIAL: NCT05922696
Title: Impact of Cholecalciferol Supplementation in Hemodialysis Patients
Brief Title: Cholecalciferol Supplementation in Hemodialysis Patients
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mona AlShahawey Ghazy, PhD, Assistant Professor of Clinical Pharmacy, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 152
Record Dates: First submitted 2023-06-20; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Anemia; Hemodialysis Complication; Vitamin D Deficiency
MeSH Terms: conditions — Anemia; Vitamin D Deficiency | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Group A: Weekly Cholecalciferol: 25 eligible hemodialysis patients on oral cholecalciferol 50.000IU Cholecalciferol, once weekly, for 3 months' duration
  Interventions: Drug: Cholecalciferol
- Group B (Active Comparator): Group b: Monthly Cholecalciferol: 25 eligible hemodialysis patients on oral cholecalciferol 200.00IU Cholecalciferol, once monthly, for 3 months' duration
  Interventions: Drug: Cholecalciferol

INTERVENTIONS:
Drug: Cholecalciferol — 50.000IU weekly in Group A , or 200.000IU monthly in Group B
  Other Names: Vitamin D3

SUMMARY:
This is prospective single-blind randomized study, in Ain Shams University hospital) in Egypt, to assess the impact of Cholecalciferol on Anemia status in regular hemodialysis outpatients

DETAILED DESCRIPTION:
This Srudy is to assess the Impact of Cholecalciferol on Anemia status in regular hemodialysis outpatients in terms of increase of Hgb >11 g/dl, transferrin saturation (TSAT) of ≥ 30%, and ferritin levels to achieve a range of (300 to < 800 ng/ml), and effect on Epoetin Dose needed. This study is also to adress the factors affecting the correcetion of Anemia by Cholecalciferol supplementation, such as oxidative stress and Inflammatory markers.

ELIGIBILITY:
Inclusion Criteria:

* : Male or female patients who are willing to participate in the trial should have been on maintenance hemodialysis sessions for not less than 3 months, aged between 18-70 years old, clinically stable (no prior hospitalization on the past three months), with serum 25(OH)D levels of less than 30 ng/ml and their iPTH levels of 150-800 pg/ml, and hemoglobin levels of less than 11 mg/dl.

Exclusion Criteria:

* Patients with previous or known hypersensitivity to cholecalciferol,
* Patients who are already on cholecalciferol therapy, or patients on immunosuppressants.
* Blood transfusion in the past 4 month, and patients who had anemia for other than renal causes,
* Those who were participating in another clinical trial within the past 4 weeks or pregnant/breastfeeding female patients were excluded as well.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-05-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
Increase serum 25-hydroxy vitamin D (25(OH)D) level to ≥ 30ng/ml | 3 months

SECONDARY OUTCOMES:
Increase in hemoglobin (Hgb) levels (11-13 mg/dl), | 3 months
TSAT levels to be ≥ 30% | 3 months
Ferritin levels to be > 300 ng/ml, but not exceeding 800 ng/ml | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt